CLINICAL TRIAL: NCT03986177
Title: Implementation of a Community Intervention to Improve Asthma Self-Management Practices in Peru
Brief Title: Asthma Implementation Research Trial
Acronym: AIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Asociacion Benefica Prisma (Other); Hospital Nacional Cayetano Heredia (Unknown); American Thoracic Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB00170462
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Asthma; Asthma in Children
Keywords: Implementation Science; Global Health; Peru
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm will receive a multi-faceted self-management intervention package.
  Interventions: Behavioral: Self-management Intervention Package
- Enhanced care (No Intervention): The control arm will receive usual care plus basic asthma education from a trained nurse educator.

INTERVENTIONS:
Behavioral: Self-management Intervention Package — Children will receive basic asthma education, based on the National Heart, Lung, and Blood Institute "A Breath of Life" asthma education program. Children/caregivers in the intervention arm will also be assigned a designated nurse case manager who will provide home visits and be available via text message and phone-based support throughout follow-up. Intervention components:
  * Interactive education and support on use of an asthma action plan
  * Locally adapted patient-provider communication tool
  * Child-oriented educational materials in comic book format
  * Modeling and hands-on practice of inhaler technique (written instructions, in person, video)
  * Education regarding environmental trigger abatement
  * Patient navigation, home visits, and goal setting support from nurse manager
  Arms: Intervention

SUMMARY:
Asthma is the most common chronic disease among children worldwide, with 80% of asthma related deaths occurring in low- and middle-income countries (LMICs), such as Peru. While evidence-based guidelines exist for asthma treatment and management, adherence to guideline-based practices is low in high-income country (HIC) and LMIC settings alike. There a clear need for effective, locally-tailored solutions to address the asthma treatment gap in low-income communities in LMICs, such as Peru. This study aims to develop and test a locally-adapted intervention package to improve adoption of self-management practices and utilization of preventive health services for asthma among children in Lima. There is a paucity of research regarding the development and testing of interventions to improve asthma self-management in LMIC settings, which experience unique or exacerbated barriers to receiving evidence-based care. To the investigators' knowledge, no studies have systematically developed and evaluated an asthma management program in Peru. Therefore, the long-term goal of this study is to disseminate locally appropriate asthma management strategies to reduce asthma-related emergency department visits and improve service utilization in LMIC settings. For the current study, the investigators will carry out a randomized controlled trial to test the effectiveness of the intervention package in a group of 110 children with asthma who will be randomized to the intervention (55 children) or no intervention (55 children) arm. Participants in the intervention group will receive case management from a designated nurse manager, who will provide ongoing educational, social, and self-management support during monthly follow-up home visits and text-message based communication. Participants will be followed up every month for data collection over a six-month period. Throughout the follow-up period, the investigators will collect data on asthma control, healthcare utilization, medication adherence, quality of life of children with asthma and the children's caregivers, caregiver mental health, fidelity to the intervention, and acceptability and feasibility. Ultimately, this study will inform the scientific community about effective strategies and treatment programs for asthma in low-income settings.

ELIGIBILITY:
Inclusion Criteria:

* Currently living in Lima, Peru
* 5-17 years of age
* Has a physician diagnosis of asthma
* Has attended the emergency room or urgent care for asthma, or has been hospitalized for asthma at least once in the previous 12 months

Exclusion Criteria:

* Family plans to move out of the study community within the next 12 months
* Co-occurring chronic respiratory or cardiovascular disorders other than asthma
* Active tuberculosis or are currently taking tuberculosis medications
* Diagnosis of HIV/AIDS

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Asthma Control as assessed by Childhood Asthma Control Test (cACT) Score | Baseline, then monthly up to 6 months
  cACT (5-11 years of age) will be administered at baseline and monthly during the follow-up period. The cACT is scored by summing the scores for all items. Overall scores ranges from 0 to 27. Lower scores indicate poorer asthma control and higher scores indicate better asthma control. Scores 19 and below suggest impaired asthma control.
Change in Asthma Control as assessed by Asthma Control Test (ACT) Score | Baseline, then monthly up to 6 months
  ACT (12-17 years of age) will be administered at baseline and monthly during the follow-up period. The ACT is scored by summing the scores for all items. Overall score ranges from 5 to 25. Lower scores indicate poorer asthma control and higher scores indicate better asthma control. Scores 19 and below suggest impaired asthma control.
Number of participants with at least one asthma-related ED or urgent care visit during the six-month follow-up period | 6 months
  Number with asthma-related emergency department (ED) or urgent care visits will be used to assess healthcare utilization.

SECONDARY OUTCOMES:
Change in Adherence to Refills and Medications Scale-7 (ARMS-7) score | Baseline, then monthly up to 6 months
  ARMS-7 will administered at baseline and monthly during the follow-up period. Score is calculated by summing the scores for all items. Overall score ranges between 7 and 28. Lower scores indicate better adherence.
Medication adherence as assessed by Dose counter-measured medication use | 6 months
  Number of puffs used divided by the number of puffs indicated to be used over monthly follow-up period.
Quality of life as assessed by Pediatric Asthma Quality of Life Questionnaire (PAQLQ)-Mini | 6 months
  Measures disease-specific quality of life in children and adolescents with asthma. The PAQLQ-mini has 13 items, each scored on a 7-point Likert scale with "1" indicating severe impairment and "7" indicating no impairment. Score is calculated by taking the average of scores for each item. Higher scores indicate better quality of life. Range: [1 to 7].
Quality of life in caregivers of children and adolescents with asthma as assessed by Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ) | 6 months
  Measures quality of life in caregivers of children and adolescents with asthma. The PACQLQ has 13 items, each scored on a 7-point Likert scale with "1" indicating severe impairment and "7" indicating no impairment. Score is calculated by taking the average of scores for each item. Higher scores indicate better quality of life. Range: [1 to 7].
Depression as assessed by Patient Health Questionnaire-9 (PHQ-9) | 6 months
  Measures depressive symptoms. Will be administered to caregivers of children and adolescents with asthma. The PHQ-9 has nine items, each scored on a Likert scale from 0 to 3. Higher scores indicate more evidence of depressive disorder of greater severity of disorder. Scores are calculated by summing the scores for all items. Range: [0 to 27].
Number of participants with asthma-related hospitalizations | 6 months
  Count of participants (children) with at least one asthma-related hospitalization during six-month follow-up period.
Number of participants with all-cause emergency department (ED) or urgent care visits | 6 months
  Count of participants with at least one all-cause ED or urgent care visit during the six-month follow-up period.
Number of participants who attend two or more outpatient appointments with healthcare provider for asthma. | 6 months
  Count of participants who attend two or more outpatient appointments with healthcare provider for asthma over six-month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Pollard, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Hospital Nacional Cayetano Heredia, Lima, Peru

REFERENCES:
- [Derived] Zevallos-Morales A, Romani-Huacani E, Psoter KJ, Flores-Flores O, Reif D, Siddharthan T, Portell M, Anguera MT, Underhill LJ, Pollard SL. Effectiveness and implementation of a multi-faceted intervention to facilitate adoption of asthma self-management practices in Peruvian children and adolescents: a hybrid type 2 individually randomized controlled trial. Front Public Health. 2026 Jan 13;13:1710746. doi: 10.3389/fpubh.2025.1710746. eCollection 2025. PMID 41607915
- [Derived] Romani ED, Siddharthan T, Lovaton N, Alvitez-Luna CC, Flores-Flores O, Pollard SL. Implementation of an intervention to improve the adoption of asthma self-management practices in Peru: Asthma Implementation Research (AIRE) randomized trial study protocol. Trials. 2020 May 4;21(1):377. doi: 10.1186/s13063-020-4207-5. PMID 32366314